CLINICAL TRIAL: NCT04768985
Title: A Phase I, Open-Label, Randomized, 2-Treatment, 2-Period, Crossover Study in Healthy Subjects to Assess the Bioequivalence of Acalabrutinib Tablet and Acalabrutinib Capsule
Brief Title: Study to Assess the Bioequivalence of Acalabrutinib Tablet and Acalabrutinib Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D8223C00013
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-03

CONDITIONS: Bioequivalence
Keywords: Pharmacokinetics; Healthy participants; Bruton tyrosine kinase; Acalabrutinib
MeSH Terms: interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment sequence 1: Treatment AB (Experimental): Participants will be randomized to receive one of the two different treatment sequences. In each treatment sequence participant will receive fixed single doses of 100 mg acalabrutinib orally (Treatment A; Treatment B) in 2 treatment periods, under fasted conditions. Treatment A will include acalabrutinib tablet and Treatment B will include acalabrutinib capsule.
  Interventions: Drug: Treatment A: Acalabrutinib tablet; Drug: Treatment B: Acalabrutinib capsule
- Treament sequence 2: Treatment BA (Experimental): Participants will be randomized to receive one of the two different treatment sequences. In each treatment sequence participant will receive fixed single doses of 100 mg acalabrutinib orally (Treatment B; Treatment A) in 2 treatment periods, under fasted conditions. Treatment A will include acalabrutinib tablet and Treatment B will include acalabrutinib capsule.
  Interventions: Drug: Treatment A: Acalabrutinib tablet; Drug: Treatment B: Acalabrutinib capsule

INTERVENTIONS:
Drug: Treatment A: Acalabrutinib tablet — Participants will receive fixed single doses of acalabrutinib tablet in 2 treatment periods, under fasted conditions.
  Other Names: CALQUENCE
Drug: Treatment B: Acalabrutinib capsule — Participants will receive fixed single doses of acalabrutinib capsule in 2 treatment periods, under fasted conditions.
  Other Names: CALQUENCE

SUMMARY:
This study is a multicenter, Phase I, open-label, randomized, 2-sequence, 2-treatment, 2-period, crossover, bioequivalence study with single doses of acalabrutinib administered orally in healthy participants. The study is designed to demonstrate the bioequivalence of acalabrutinib tablet (Treatment A) compared with marketed acalabrutinib capsule (Treatment B) in the fasted state.

DETAILED DESCRIPTION:
Eligible healthy participants will be randomized to receive either treatment sequence 1 (AB) or treatment sequence 2 (BA), as follows:

* Treatment A: Acalabrutinib tablet, 100 mg, fasted state
* Treatment B: Acalabrutinib capsule, 100 mg, fasted state

Participants will receive fixed single doses of acalabrutinib on 2 occasions, under fasted conditions.

The study will comprise:

* Visit 1: A screening period of up to 28 days before first dosing.
* Visit 2: Two treatment periods:

  * Participants will be admitted to the study center on Day -2 of Treatment Period 1 to confirm eligibility before first dosing. Eligibility criteria will be reconfirmed on Day -1 of each treatment period.
  * On Day 1 of Treatment Periods 1 and 2, participants will be administered the assigned treatment (A or B) as randomized, followed by a protocol defined washout period between Treatment Periods 1 and 2.
* Visit 3: A Follow-up Visit/Early Termination Visit at 7 to 10 days after last administration of study drug.

Each participant will be involved in the study for approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females must have a negative pregnancy test at Screening and on admission to the study center, must not be lactating, and must be of non-childbearing potential, confirmed at Screening, by fulfilling protocol defined criteria
* Have a body mass index between 18.5 and 30 kg/m^2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive, at Screening
* Non-smokers and those participants who have not smoked (including e cigarettes) or used nicotine products (cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or any other nicotine containing products) within the 90 days prior to Screening
* Calculated creatinine clearance (CrCl) ≥ 90 mL/min as determined by Cockcroft-Gault method (using actual body weight)

Males:

CrCl = Weight (kg) × (140 - Age)/72 × serum creatinine (mg/dL) in mL/min

Females:

CrCl = Weight (kg) × (140 - Age) × 0.85/72 × serum creatinine (mg/dL) in (mL/min)

Exclusion Criteria:

* History or presence of any clinically significant disease (including active coronavirus disease 2019 [COVID-19] infection) or disorder
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any clinically significant illness, medical/surgical procedure, or trauma within 30 days of the first administration of study drug
* Any clinically significant abnormalities in hematology, coagulation, clinical chemistry, or urinalysis results, at Screening and prior to first dose, as judged by the Investigator and defined as:

  (i) Hemoglobin less than lower limit of normal (ii) Absolute neutrophils less than lower limit of normal (iii) Platelets less than lower limit of normal (iv) Serum alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase or serum bilirubin (total bilirubin and direct bilirubin) > upper limit of normal
* Any clinically significant abnormal findings in vital signs at Screening or on Day 1 (eg, systolic BP < 90 mmHg or > 140 mmHg; diastolic BP < 50 mmHg or > 90 mmHg; pulse < 45 or > 90 bpm)
* Any clinically significant abnormalities on standard 12-lead ECG at Screening or on Day 1
* Any positive result for HBsAg, hepatitis C antibody, and HIV testing, at Screening
* Has received a new chemical entity (defined as a compound which has not been approved for marketing) within 90 days of the first administration of study drug in this study. The period of exclusion begins 90 days after the final dose or 30 days after the last visit whichever is the longest
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to acalabrutinib
* Positive screen for drugs of abuse or cotinine and alcohol, at Screening and on admission to the study center
* Treatment with prescription or non-prescription drugs or other products known to be strong CYP3A, P-gp, or breast cancer resistance protein (BCRP) inhibitors or substrates of BCRP or MATE1 (within 14 days before first administration of study drug or longer if the medication has a long half life) and strong CYP3A inducers (within 28 days before first administration of study drug or longer if the medication has a long half life)
* Use of any prescribed or non prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose), and minerals during the 14 days prior to the first administration of study drug or longer if the medication has a long half life
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) as judged by the Investigator
* Inability to swallow acalabrutinib tablets or acalabrutinib capsules
* Evidence of ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections)
* Participant has a positive test result for severe acute respiratory syndrome coronavirus 2 reverse transcriptase polymerase chain reaction before randomization
* Participant has clinical signs and symptoms consistent with COVID-19, eg, fever, dry cough, dyspnea, sore throat, fatigue, or confirmed infection by appropriate laboratory test within the last 4 weeks prior to Screening or on admission
* History of severe COVID-19 (hospitalization, extracorporeal membrane oxygenation, mechanically ventilated)
* Participants who are regularly exposed to COVID-19 as part of their daily life (eg, health care professionals working in COVID-19 wards or at emergency departments)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve from zero to infinity (AUCinf) of Acalabrutinib | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the AUCinf of acalabrutinib capsule with the tablet.
Area under the plasma concentration time curve from zero to the last quantifiable concentration (AUClast) of Acalabrutinib | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the AUClast of acalabrutinib capsule with the tablet.
Maximum observed plasma (peak) drug concentration (Cmax) of Acalabrutinib | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the Cmax of acalabrutinib capsule with the tablet

SECONDARY OUTCOMES:
Area under plasma concentration time curve from zero to infinity (AUCinf) of ACP-5862 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the AUCinf of acalabrutinib capsule with the tablet.
Area under the plasma concentration time curve from zero to the last quantifiable concentration (AUClast) of ACP-5862 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the AUClast of acalabrutinib capsule with the tablet.
Maximum observed plasma (peak) drug concentration (Cmax) of ACP-5862 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the Cmax of acalabrutinib capsule with the tablet.
Time to reach peak or maximum concentration (tmax) following drug administration for acalabrutinib and ACP-5862 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the tmax of acalabrutinib capsule with the acalabrutinib tablet.
Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve (t½λz) for acalabrutinib and ACP-5862 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the t½λz of acalabrutinib capsule with the acalabrutinib tablet.
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRT) for acalabrutinib and ACP-5862 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the MRT of acalabrutinib capsule with the acalabrutinib tablet.
Terminal rate constant, estimated by log linear least squares regression of the terminal part of the concentration time curve (λz) for acalabrutinib and ACP-5862 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the λz of acalabrutinib capsule with the acalabrutinib tablet.
Metabolite (ACP-5862) to parent (acalabrutinib) ratio based on AUCinf and/or AUClast (M:P[AUC]) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the M:P[AUC] of acalabrutinib capsule with the tablet.
Metabolite (ACP-5862) to parent (acalabrutinib) ratio based on Cmax (M:P [Cmax]) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose
  To compare the M:P[Cmax] of acalabrutinib capsule with the tablet.
Number of participants with adverse events and serious adverse events | From screening day (Day -28) until Follow-up/end of treatment visit (at 7 to 10 days after last study drug administration)
  Comparison of the safety and tolerability of single doses of acalabrutinib capsule with the tablet.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — Parexel Early Phase Clinical Unit Baltimore Harbor Hospital 3001 South Hanover St. Baltimore, MD 21225 USA
Locations (3):
- United States (3):
  - Research Site, Glendale, California
  - Research Site, Brooklyn, Maryland
  - Research Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search